CLINICAL TRIAL: NCT04002206
Title: Immediate Effects of Post-isometric Relaxation and Static Stretching on Quadriceps Muscle During Vertical Jump in Volley Ball and Basketball Players
Brief Title: Comparison of Muscle Energy Technique vs Static Stretch in Vertical Jump of Basketball and Volleyball Player
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Riphah IU M Faheem Afzal
Record Dates: First submitted 2019-06-11; First posted 2019-06-28 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Healthy
Keywords: Muscle Energy Technique; Post isometric relaxation technique.

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique (Experimental): Post isometric relaxation technique was used in experimental group
  Interventions: Other: Muscle Energy Technique
- Static Stretch (Active Comparator): Static stretching was given in control group
  Interventions: Other: Static Stretch

INTERVENTIONS:
Other: Muscle Energy Technique — In experimental group, post-isometric relaxation technique has given to the athletes. The position of athlete was prone and the involved group of muscle was quadriceps. Firstly end range of the quadriceps muscle group assess and guide the athlete to put 20% of their maximum voluntary contraction and physiotherapist resist the athlete and isometric contraction of quadriceps remain for 6-10 seconds
  Arms: Muscle Energy Technique
Other: Static Stretch — Control group has treated with static stretching after the pre-assessment that includes three repetitions with duration of fifteen seconds with twenty second rest intervals on lower extremities
  Arms: Static Stretch

SUMMARY:
A randomized control trial study was conducted in Islamic International University Islamabad from 1st August 2017 to 31st January 2018 according to the set criteria. A total number of 29 athletes age between 18-35 and playing as part time/ domestic level included in this study. Data were divided into experimental group (n=15) and control group (n=14) by random sampling technique. Post isometric relaxation technique was used in experimental group and static stretching was given in control group. Baseline reading was taken before intervention and post intervention reading taken immediately after application of intervention. Data analyzed through SPSS 20.

DETAILED DESCRIPTION:
Vertical jump is defined as the ability of athlete to elevate off the ground from standstill.There are two types of vertical jump which re squat vertical jump and vertical stop jump. There was a strong correlation between maximal strength in half squats and sprint performance and jumping height.

Muscle energy technique(METS) is the procedure which involves voluntary contraction of muscle in specific direction with different angles against a counterforce applied by clincian.METS is used to enhance strength of group of muscle, increase afferent input to facilitate reflexive stabilization and increase endurance in coordinated movement patterns.

Athletes perform dynamic stretching before sports involvement. Study shows that three 30 seconds stretch enhance muscle length immediatley after stretching.

A study conducted in 2003 to see the effects of muscle energy technique on hamstring extensibility, the conclusion of this study that muscle energy technique produced an immediate increase in passive knee extension.

A study conducted on immediate effect of two muscle energy techniques on quadriceps muscle during vertical jump. The study suggests concentric muscle energy technique on quadriceps muscle is the most appropriate technique to potentiate height jump performance and stretch-shorten cycle function in counter-movement jump.

Athletes ususully perfrom stretching exercises in warm up before involvement to sports.Study suggest that dynamic stretching is more suitable for use as part of warmup in young athletes. Athletes invlve in high intensity exercise demand stretch shorten cycle, stretching may be important for injury prevention. Stretching also reduce the peak torque and mean power output.

ELIGIBILITY:
Inclusion Criteria:

* Athletes (volley ball and basketball players) playing at part time/domestic level.
* Athletes age between 18-35 Years.

Exclusion Criteria:

* Athletes having history of sprain or strain in lower limbs within last 6 months.
* Athletes having any neuro-musculoskeletal, cardiovascular pathology

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Due to limitation in sports club
Enrollment: 29 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Vertical Jump - Force Plates | Day 1
  Athletes starting position is squat position (Which is the baseline position) on the force-plates and did jump by saying jump, then Jump and sway were noted by physical therapist in seconds
Muscle Recruitment: through Electromyography | Day 1
  During vertical jump athletes quadriceps muscle recruitment is noted by noting the amplitude
30 Meter sprint | Day 1
  Athletes start its 30 meter sprint with maximum speed and it is used to check the maximum strength in seconds
Ground Reaction force (flight time):- through Force plates | Day 1
  Athletes starting position is squat position on the force-plates and did jump by saying jump and the flight time were noted by physical therapist in newton

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PHD, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wisloff U, Castagna C, Helgerud J, Jones R, Hoff J. Strong correlation of maximal squat strength with sprint performance and vertical jump height in elite soccer players. Br J Sports Med. 2004 Jun;38(3):285-8. doi: 10.1136/bjsm.2002.002071. PMID 15155427
- [Background] de Weijer VC, Gorniak GC, Shamus E. The effect of static stretch and warm-up exercise on hamstring length over the course of 24 hours. J Orthop Sports Phys Ther. 2003 Dec;33(12):727-33. doi: 10.2519/jospt.2003.33.12.727. PMID 14743986
- [Background] Ballantyne F, Fryer G, McLaughlin P. The effect of muscle energy technique on hamstring extensibility: the mechanism of altered flexibility. Journal of Osteopathic Medicine. 2003 Oct 1;6(2):59-63
- [Background] 4. Gentil-Bécoz J, Royal S, Locatelli M, Perez GM. The immediate effects of two muscle energy techniques on quadriceps muscle during vertical jumps: A pilot Study. Journal of Bodywork and Movement Therapies. 2015 Oct 1;19(4):672-3
- [Background] Carvalho FL, Carvalho MC, Simao R, Gomes TM, Costa PB, Neto LB, Carvalho RL, Dantas EH. Acute effects of a warm-up including active, passive, and dynamic stretching on vertical jump performance. J Strength Cond Res. 2012 Sep;26(9):2447-52. doi: 10.1519/JSC.0b013e31823f2b36. PMID 22067244
- [Background] Witvrouw E, Mahieu N, Danneels L, McNair P. Stretching and injury prevention: an obscure relationship. Sports Med. 2004;34(7):443-9. doi: 10.2165/00007256-200434070-00003. PMID 15233597
- [Background] Cramer JT, Housh TJ, Weir JP, Johnson GO, Coburn JW, Beck TW. The acute effects of static stretching on peak torque, mean power output, electromyography, and mechanomyography. Eur J Appl Physiol. 2005 Mar;93(5-6):530-9. doi: 10.1007/s00421-004-1199-x. Epub 2004 Dec 15. PMID 15599756